CLINICAL TRIAL: NCT06044571
Title: Optimizing Telehealth-delivery of a Weight Loss Intervention in Older Adults With Multiple Chronic Conditions: A Sequential, Multiple Assignment, Randomized Trial
Brief Title: Optimizing Telehealth-delivery of a Weight Loss Intervention in Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 23-1146; 1R01AG077163-01A1 (NIH)
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Obesity; Multiple Chronic Conditions
MeSH Terms: conditions — Obesity; Multiple Chronic Conditions | interventions — Directive Counseling

STUDY DESIGN:
Intervention Model Description: A single site two-stage, Phase III clinical trial using a SMART design, will assess the superiority between two first-line strategies (prescriptive, behavioral) on percent weight loss at 52 weeks
Who Masked: Participant, Care Provider
Masking Description: This trial will have a single-masked design, so the team assessing study outcomes is masked to intervention assignment. Participants will be asked not to reveal their assignment. Arm assignment cannot be blinded due to the study's design. The assessment team will schedule assessments to minimize contact with the intervention team to maintain separation. Data entry and analysis will be blinded to the study investigators, besides Kosorok and team. Assessments will be done at different times and in separate areas at the study site. The intervention setting for participants will be in their homes. To enhance continued masking, participants will be asked not to disclose their assigned group and not to discuss their intervention arms during assessment sessions. Assessment of compliance to the intervention will be performed by the intervention team and not by the outcome assessment team. The investigators will be blinded to data analysis, collection, and study arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Prescriptive (Active Comparator): A diet and exercise prescription individually tailored to each participant's multiple chronic health conditions will provide concrete advice with less autonomy, and will minimize risks of physiologic changes due to weight loss (hypoglycemia, hypotension, muscle loss). Licensed, trained professionals- Registered Dietician Nutritionists (RDNs) and Physical Therapists (PTs) will introduce clinical reasoning, knowledge, and experience, assess biological adaptations to weight loss, modify prescriptions based on changing medical needs, and provide real-time and asynchronous guidance. Registered Dietician Nutritionists (RDNs) and Physical Therapists (PTs) will deliver group and individual, live sessions to the home by telemedicine. Sessions will last 60-min (Registered Dietician Nutritionist: 20 min; Physical Therapy: 40 min).
  Interventions: Other: Prescriptive
- Behavioral (Active Comparator): Health coaches have a bachelor's degree and take a 6-8-week certification program. Health coaches will use a structured manual involving evidence-based behavior change techniques (problem-solving, self-regulation, motivation). Group and individual sessions will be via telemedicine.
  Conceptual model targets include:
  1. barrier identification: problem-solving to identify and address barriers to meet goals
  2. self-regulation: a focus on self-monitoring and behavior goals with feedback
  3. autonomous motivation: self-selecting goals, motivational interviewing use, and creating plans; and (d) self-efficacy: learning from group experiences, verbal persuasion, and encouraging pursuit of goals in the face of setbacks.
  Interventions: Behavioral: Behavioral
- Responders to Prescriptive- Continue Prescriptive (Experimental): The prescriptive strategy will continue among participants who responded to this intervention well initially, meaning that participants who lost greater than or equal to 2.5 percent (%) of their body weight using the prescriptive intervention. Participants will continue their diet and exercise programs that were initially tailored to them.
  Interventions: Other: Prescriptive
- Non-responders to Prescriptive- Switch to Behavioral (Experimental): Participants who lost less than 2.5 percent (%) of their body weight initially will be randomized to a different type of intervention. One possibility could be that participants switch first-line treatment from a prescriptive strategy to the alternative (behavioral) as participants may need motivation or problem-solving.
  Interventions: Behavioral: Behavioral
- Non-responders to Prescriptive- Combination of Prescriptive and Behavioral (Experimental): Participants who lost less than 2.5 percent (%) of their body weight early on will be re-randomized to a different type of intervention. One possibility could be that participants will have a combined prescriptive and behavioral intervention- three guideline-advised strategies that may be synergistic in a subset of participants requiring knowledge, and needing goal setting and problem-solving skills. This approach is available in multispecialty, tertiary care obesity clinics.
  Interventions: Other: Prescriptive; Behavioral: Behavioral
- Responders to Behavioral- Continue Behavioral (Experimental): The behavioral strategy will continue among participants who responded to this intervention well initially, meaning that participants who lost greater than or equal to 2.5 percent (%) of their body weight using the behavioral intervention.
  Interventions: Behavioral: Behavioral
- Non-responders to Behavioral- Switch to Prescriptive (Experimental): Participants who lost less than 2.5 percent (%) of their body weight early on will be re-randomized to a different type of intervention. One possibility could be that participants switch first-line treatment strategy to the alternative (prescriptive) as participants may need knowledge to support adherence.
  Interventions: Other: Prescriptive
- Non-responders to Behavioral- Combination of Prescriptive and Behavioral (Experimental): Participants who lost less than 2.5 percent (%) of their body weight early on will be re-randomized to a different type of intervention. One possibility could be that participants will have a combined prescriptive and behavioral intervention - three guideline-advised strategies that may be synergistic in a subset of participants requiring knowledge, and needing goal setting and problem-solving skills. This approach is available in multispecialty, tertiary care obesity clinics.
  Interventions: Other: Prescriptive; Behavioral: Behavioral

INTERVENTIONS:
Other: Prescriptive — Prescriptive A diet and exercise prescription individually tailored to each participant's multiple chronic health conditions will provide concrete advice with less autonomy, and will minimize risks of physiologic changes due to weight loss (hypoglycemia, hypotension, muscle loss). Licensed, trained professionals, Registered Dietician Nutritionists (RDNs) and Physical Therapists (PTs), will introduce clinical reasoning, knowledge, and experience, assess biological adaptations to weight loss, modify prescriptions based on changing medical needs, and provide real-time and asynchronous guidance. Registered Dietician Nutritionists (RDNs) and Physical Therapists (PTs)will deliver group and individual, live sessions to the home by telemedicine. Sessions will last 60-min (Registered Dietician Nutritionist: 20 min; Physical Therapist: 40 min).
  Arms: Non-responders to Behavioral- Combination of Prescriptive and Behavioral; Non-responders to Behavioral- Switch to Prescriptive; Non-responders to Prescriptive- Combination of Prescriptive and Behavioral; Prescriptive; Responders to Prescriptive- Continue Prescriptive
Behavioral: Behavioral — Behavioral Health coaches have a bachelor's degree and take a 6-8-week certification program. Behavioral Health coaches will use a structured manual involving evidence-based behavior change techniques (problem-solving, self-regulation, motivation). Group and individual sessions will be via telemedicine.
  Arms: Behavioral; Non-responders to Behavioral- Combination of Prescriptive and Behavioral; Non-responders to Prescriptive- Combination of Prescriptive and Behavioral; Non-responders to Prescriptive- Switch to Behavioral; Responders to Behavioral- Continue Behavioral

SUMMARY:
This study seeks to answer the fundamental questions of which initial, first-line weight loss intervention should be offered to older adults with obesity and multiple chronic conditions and how to address the high non-response rates observed with most conventional strategies. A sequential, multiple assignment, randomized trial (SMART) design will permit the evaluation of treatment combinations that maximize weight loss and will provide data on constructing a future tailored, adaptive intervention. If successful, these findings will identify interventions that could markedly improve health and quality of life of these older adults, reduce long-term disability, and lower healthcare costs

DETAILED DESCRIPTION:
Purpose: Consistent with the research priorities of the National Institute on Aging, this research protocol will investigate the optimal intervention sequence to achieve weight loss in older adults with obesity and more than 2 chronic conditions, termed multiple chronic conditions (MCC). To this end, the specific aims are to: 1) test the superiority of an initial prescriptive or behavioral intervention using an adaptive strategy for early non-responders; 2) assess the patterns of initial weight loss and compare strategies for non-responders using an adaptive strategy; and 3) examine the cost-effectiveness from a societal perspective for maintaining weight loss of the proposed sequences at 52 weeks.

Procedures (methods): The investigators will conduct a 52-week, two-stage, Sequential, Multiple Assignment, Randomized Trial (SMART) enrolling 180 older adults with obesity and MCC to compare two weight loss interventions: 1) a prescriptively-focused, medically-tailored, weight loss intervention (prescriptive), or 2) a behaviorally-focused, health coaching intervention (behavioral). Consistent with a SMART design, at 8 weeks, the investigators will randomize early non-responders (weight loss of < 2.5%) to (a) a combination of prescriptive and behavioral interventions; or (b) switching to either a prescriptive, medically-tailored model (or vice versa).

Aim 1 - Efficacy Test the superiority of an initial prescriptive vs. behavioral intervention on the differences in weight loss (primary outcome) and secondary outcomes, using an adaptive strategy for early non-responders in a 52-week, telehealth-based SMART. At 52-weeks, percent weight loss (primary outcome) will be greater among patients initially randomized to a prescriptive intervention, as will global health and physical function, anthropometry, behavioral treatment targets and risk factors, and clinical indices (secondary outcomes).

Aim 2 - Precision Medicine Assess the patterns of initial weight loss and compare strategies for non-responders to weight loss (combined prescriptive and behavioral, or switching initial treatment strategies [prescriptive to behavioral, or behavioral to prescriptive]). The investigators will estimate an adaptive strategy (dynamic treatment regime) to give the right intervention to the right participant. The investigators hypothesize that this dynamic regime will lead to a better outcome, on average, compared to the best non-adaptive (fixed) regime

Aim 3 - Cost-Effectiveness Examine the cost-effectiveness from a societal perspective at 52-weeks. For the initial, first-line interventions, the investigators will estimate the incremental cost per percent weight change and assess secondary outcomes of the incremental cost for maintaining at least a 5% weight loss, and quality-adjusted life years. The investigators will also model the cost-effectiveness of the precision medicine approach predicted to have the greatest individualized likelihood of weight loss response.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria based on chart review at the time of screening (within 8 weeks of randomization):

* Community-dwelling adult living independently (not a resident of a nursing home or an assisted living);
* Aged 65-85 years (unclear benefits of weight loss if >85 years)
* Obesity (body mass index: ≥30 kg/m2);
* English-speaking;

  -≥2 chronic medical conditions that require ongoing care (excluding dementia and osteoporosis as a chronic condition) - these are based on Medicare' MCC (e.g., alcohol abuse, arthritis (osteoarthritis, rheumatoid), asthma, atrial fibrillation, autism spectrum disorders, cancer (breast, colorectal, lung, prostate), chronic kidney disease, chronic obstructive pulmonary disease, depression, diabetes, drug/substance abuse, heart failure, hepatitis, Human Immunodeficiency Virus / Acquired Immunodeficiency Disease Syndrome, hyperlipidemia, hypertension, ischemic heart disease, schizophrenia/other psychotic disorders, stroke). We acknowledge that there are no fully defined definitions and hence we will be assessing MCC (or multimorbidity) in different manners;
* medical clearance by PCP (Primary Care Provider)
* Callahan cognitive screen ≥ 3 correct items; items (a score of three or more correct items indicates an ability to consent);
* OARS (Older Americans Resources and Services)survey score of ≥12; (a score of 12 or more indicates no impairments or disability)
* Readiness to change score of ≥6/10;

Exclusion Criteria:

Any individual who meets one or more of the following criteria will be excluded from participation based on chart review at the time of screening (within 8 weeks of randomization):

* documented diagnosis in the electronic health record of dementia of any type;
* documented diagnosis in the electronic health record of weight loss surgery in the past;
* untreated psychiatric disorder that would impair the ability to participate (bipolar, schizophrenia) based on medical record review;
* life-threatening illness;
* terminal illness (e.g., palliative care, hospice patient) based on medical record review whose life expectancy is <12 months as determined by a physician;
* nursing home or hospital admission in past three months;
* advanced comorbidities based on medical record review;
* heart - recent hospital admission for heart failure, myocardial infarction, stroke in past 3 months, unstable disease (new york class III or IV congestive heart failure);
* chronic renal failure - chronic kidney disease stage IV or V (e.g., GFR [glomerular filtration rate] <30ml/min);
* non-skin cancer - history of requiring active treatment in the past year;
* liver failure or cirrhosis;
* chronic obstructive pulmonary disease - on oxygen or requiring steroids;
* weight loss contraindication as noted by the PCP;
* instability of weight loss, which is greater than 5% weight loss in the past 12 weeks;
* anti-obesity medications including orlistat, semaglutide, liraglutide, tirzepetide, naltrexone-bupropion and phentermine prior to initiation of study procedures;
* current use of bone acting medications (e.g., raloxifene, calcitonin, parathyroid hormone during the past year, Parathyroid Hormone Analogues (PTH-analogues [e.g., teriparatide, abaloparatide], sclerostin) inhibitors (romosozumbab), RANK ligand inhibitors (denosumab) or bisphosphonates during the last two years;
* osteoporosis by medical record (t-score -2.5 and below on hip or spine scan) or history of fragility fractures;
* elective surgery in next 12 months;
* recent (<1 mo) COVID-19 infection;
* current or past participation (in the past 12 months) in another weight-loss study;
* Planning on moving out of the area in the next 18 months.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in weight from baseline | 8, 26, 52 weeks
  Absolute change in weight percentage (%) over time from baseline to 52-weeks. Weight will be objectively measured on a digital scale. A negative number will indicate weight loss.

SECONDARY OUTCOMES:
Change in Patient reported outcomes measurement information systems (PROMIS)- Global health | 0, 8, 16, 26, 52 weeks
  PROMIS (Patient Reported Outcomes Measurement Information System) gauges physical, mental, and social aspects of health (5-point scale). A mean standardized score for the population is 50; 10 points indicate one standard deviation. Higher scores indicate better health. Range (0-100)
Change in Patient reported outcomes measurement information systems (PROMIS)- Physical function | 0, 8, 16, 26, 52 weeks
  Self-reported physical function (5-point scale) measure that is a responsive measure evaluating mobility and activities of daily living; A mean standardized score for the population is 50; 10 points indicate one standard deviation. Higher scores indicate better health. Range (0-100)
Change in 30-second sit-to-stand from baseline | 0, 8, 26, 52 weeks
  This is a construct of physical function that predicts falls and disability and is sensitive to change. The 30-second sit-to-stand test is administered using a folding chair without arms and involves recording the number of stands from a seated position a person can complete in 30 seconds. Change in 30-s sit-to-stand in repetitions over time will be reported from baseline to 52-weeks. An improvement in repetitions will represent an improvement of physical function. The continuous value correlates with quadriceps Minimal Clinically Important Difference (2.0 repetitions)
Change in grip strength from baseline | 0, 8, 26, 52 weeks
  An objective measure that relates to upper and lower extremity strength, and predicts mobility disability. Using a Jamar dynamometer, change in participant's maximal grip strength measurement in kilograms from baseline. Absolute change in grip strength in kilograms over time will be reported from baseline to 52-weeks. An increase in kilograms represented on the device will represent an improvement of physical function. No cutoffs will be used for this - the research team will be use the continuous value.
Change in gait speed from baseline | 0, 8, 26, 52 weeks
  Gait speed (measured in meters/second or m/s) measures how long it takes a person to travel a given distance. It is A simple, clinical measure of objective physical function that reflects health and functional status and predicts falls, disability, and mortality. Gait Speed is measured using the time in seconds it takes a participant to complete a 4 meter course while walking at a usual pace. Gait speed is measured as distance (meters) ÷ time (seconds). An absolute change in gait speed will be the difference from follow-up measures and baseline. An improvement in gait speed represents an improvement in physical function. Units are meters/second. Normal >1.2m/s.
Change in 6-minute walk from baseline | 0, 8, 26, 52 weeks
  A measure of aerobic endurance (normal distance 400-700m) that is a surrogate for submaximal aerobic/cardiovascular fitness. Clinically significant change ranges between 14-30.5 m.
Change in waist circumference from baseline | 0, 8, 26, 52 weeks
  Absolute change in waist circumference in centimeters (cm) over time from baseline. Waist circumference will be measured objectively using a tape measure. A negative number will indicate a loss in waist circumference
Change in hip circumference from baseline | 0, 8, 26, 52 weeks
  Absolute change in hip circumference in centimeters (cm) over time from baseline. Hip circumference will be measured objectively using a tape measure. A negative number will indicate a loss of hip circumference
Proportion with greater than or equal to 5% weight loss | 8, 26, 52 weeks
  The proportion achieving a clinically significant 5% weight loss
Change in % body fat from baseline | 0, 26, 52 weeks
  Dual x-ray absorptiometry (General Electric Lunar iDXA) software will assess total body fat % (percent). A reduction in the percentage of total body fat is suggestive of improvements in health related outcomes.
Change in volume of visceral fat from baseline | 0, 26, 52 weeks
  Dual x-ray absorptiometry (General Electric Lunar iDXA) software will assess visceral fat mass % (percent). A reduction in visceral fat volume is suggestive of improvements in health related outcomes.
Change in appendicular lean mass from baseline | 0, 26, 52 weeks
  Dual x-ray absorptiometry (General Electric Lunar iDXA) software will assess percent (%) lean mass (total, segmental). A reduction in lean mass percentage is suggestive of worsening of health related outcomes.
Late-life function and disability instrument | 0, 8, 16, 26, 52
  Self-reported 32-item physical function measure consisting of function and life-task items that correlate with gait speed and lower-limb function. A 2-point difference is clinically significant. Range, (scaled score, 0-100). Higher scores indicate better performance and less limitation than lower scores.
Change in Pittsburgh Fatigability questionnaire | 0, 8, 16, 26, 52 weeks
  The 15-item Pittsburgh Fatigability Scale measures perceived fatigue of sedentary, social, lifestyle and physical activities (light-high intensity, 0-50 scale). Cutoff of ≥15 and ≥13 indicate higher physical and mental fatigue that may lead to reduced performance or restricted activity. Higher scores indicate greater perceived physical or mental fatigability. A reduction in the absolute change in score suggests improvements in fatigue.
Change in Self-efficacy- exercise | 0, 8, 16, 26, 52 weeks
  The Self-Efficacy for Exercise Scale (range 0-90) is based on the Social Cognitive Theory (higher scores mean higher self-efficacy for initiating/maintaining exercise). A positive change in self-efficacy reflects better outcomes, and a negative change reflects worse outcomes.
Change in Self-efficacy- nutrition | 0, 8, 16, 26, 52 weeks
  The 8-item Weight-Efficacy Lifestyle Short Form measures confidence in adopting and maintaining weight loss behaviors. A 15-point change was related to a 25% weight loss in bariatric surgery participants. Range (0-80). A positive change in self-efficacy reflects better outcomes, and a negative change reflects worse outcomes.
Change in Self-efficacy- technology | 0, 8, 16, 26, 52 weeks
  A 10-item Likert scale (1-10) will measure daily Technology Self-Efficacy (higher score means higher self-efficacy). Range (0-100)
Change in Goal setting- exercise | 0, 8, 16, 26, 52 weeks
  Only conducted in the Behavioral arms. This is a Likert Scale question, where answers can range from 1-10, with higher scores indicating better goal setting abilities
Change in Goal setting- nutrition | 0, 8, 16, 26, 52 weeks
  Only conducted in the Behavioral arms. This is a Likert Scale questionnaire, where answers can range from 1-10, with higher scores indicating better goal setting abilities.
Change in Goal setting- technology | 0, 8, 16, 26, 52 weeks
  Only conducted in the Behavioral arms. This is a Likert Scale questionnaire, where answers can range from 1-10, with higher scores indicating better goal setting abilities.
Change in social support for diet | 0, 8, 16, 26, 52 weeks
  A validated scale that assesses friends/family support for engaging in dietary changes. Higher scores indicate higher social support. Each are scored for family and friends separately (range 0-100).
Change in social support for exercise | 0, 8, 16, 26, 52 weeks
  A validated scale that assesses friends/family support for engaging in dietary exercises. Higher scores indicate higher social support. Each are scored for family and friends separately (range 0-60).
Treatment self-regulation: diet | 0, 8, 16, 26, 52 weeks
  A validated 15-item, 7-point scale (range 0-100) reflecting autonomous motivation and controlled motivation. Higher scores indicate better outcomes.
Treatment self-regulation: exercise | 0, 8, 16, 26, 52 weeks
  A validated 15-item, 7-point scale (range 0-100) reflecting autonomous motivation and controlled motivation. Higher scores indicate better outcomes.
Change in caloric intake | 0, 8, 16, 26, 52 weeks
  Using the Automated Self-Administered 24-hour Dietary Assessment (ASA-24), the investigators will measure caloric intake per day. Change measured in the difference between calories per day at baseline, throughout study, and follow-up assessment. This is an automated food recall that assess caloric intake. A change in caloric intake will be reported in kcal per day. Reduction in caloric input suggests reduced calorie intake.
Physical activity: community healthy activities model program for seniors | 0, 8, 16, 26, 52 weeks
  This questionnaire, known as CHAMPS (community healthy activities model program for seniors), will assess activity levels and types (weekly caloric expenditure; frequency of activities) and their changes. The investigators will use a standardized algorithm to assess low, moderate, vigorous activity and caloric output
Patient activation measure | 0, 8, 16, 26, 52 weeks
  Patient Activation Measure assesses knowledge, skills & confidence for managing health revealing insights into motivators, behaviors, attitudes & outcomes (4 points each; score 0-100, low to high)
Fitbit use- Wear/non-wear time | 0, 8, 16, 26, 52 weeks
  Measurement using Fitbit data of the time spent during the day wearing the device.
Fitbit use- activity/steps | 0, 8, 16, 26, 52 weeks
  Evaluation using Fitbit data of the average number of steps (and total number to that point) a participant has engaged in
Attendance | 52 weeks
  Feasibility of study procedures measured as the mean attendance rate of all participants. Participant attendance rate = (total # of visits attended / total # of visits scheduled) x 100. There are no cut-off scores for interpretation. Higher scores indicate higher feasibility
Acceptability of Study Intervention | 52 weeks
  Measured through an end of study satisfaction survey, acceptability is measured on a 10 point Likert scale conducted on all participants at 52-weeks. This is rated on a 1 (strongly disagree) to 10 (strongly agree) survey.
Percent of participants rating the intervention as acceptable | 52 weeks
  Conducted on all participants using a 1-5 Likert scale to assess appropriateness of the study intervention measures using the following: completely disagree, disagree, neither agree or disagree, agree, completely agree. Acceptability is reported as Agree or Completely Agree responses. Percent is calculated as total number of participants rating as agree or complete agree divided by the number of total participants.
Telehealth satisfaction | 52 weeks
  A end-of-study questionnaire that assesses patient satisfaction regarding the use of Telehealth (Likert scale, 1-10). Range 0-100. Higher scores indicate better outcomes.
Telehealth usability survey | 52 weeks
  A single item Likert scale (1-10) will measure usefulness, ease of use, effectiveness, reliability & satisfaction of telemedicine. This will be measured at the conclusion of the study intervention. Range 0-100. Higher scores indicate better outcomes.
Change in systolic blood pressure | 0, 8, 26, 52 weeks
  The difference between baseline and follow-up values-measured in mmHg (millimeters of mercury)- a value of 5mmHg (millimeters of mercury) is clinically significant
Change in diastolic blood pressure | 0, 8, 26, 52 weeks
  The difference between baseline and follow-up values (measured in mmHg)- a value of 5mmHg (millimeters of mercury) is clinically significant
Change in low density lipoprotein blood levels | 0, 52 weeks
  The difference between baseline and follow-up values measured in mg/dL (milligrams per deciliter) using a lipid panel. Levels >100mg/dL would be potentially clinically actionable.
Change in high density lipoprotein blood levels | 0, 52 weeks
  The difference between baseline and follow-up values measured in mg/dL (milligrams per deciliter) using a lipid panel
Change in total cholesterol blood levels | 0, 52 weeks
  The difference between baseline and follow-up values measured in mg/dL (milligrams per deciliter) using a lipid panel
Change in glucose blood levels | 0, 52 weeks
  The difference between baseline and follow-up values, units in mg/dL (milligrams per deciliter). A glucose level >126mg/dL is considered diabetic.
Change in calf circumference from baseline | 0, 8, 26, 52 weeks
  Change in calf circumference in centimeters (cm) over time from baseline to 12-weeks. Calf circumference will be measured objectively using a tape measure. A negative number will indicate a loss in calf circumference
Change in arm circumference from baseline | 0, 8, 26, 52 weeks
  Change in arm circumference in centimeters (cm) over time from baseline to 12-weeks. Arm circumference will be measured objectively using a tape measure. A negative number will indicate a loss in arm circumference.

CONTACTS AND LOCATIONS:
Overall Officials: John Batsis, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Center for Aging and Health, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No